CLINICAL TRIAL: NCT06043921
Title: Multicenter Study of Circulating Tumor DNA in Patients With Pancreatic Cancer Using a Personalized Panel
Acronym: ARTEMIS-PC
Status: Recruiting | Type: Observational
Sponsor: Invitae Corporation (Industry)
Collaborators: National Cancer Center Hospital East (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-003
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Cancer
Keywords: Circulating tumor DNA; Molecular Residual Disease; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients who have been diagnosed with pancreatic cancer and who have formalin-fixed paraffin-embedded (FFPE) tissue available will provide FFPE and whole-blood samples for the initial testing. Blood samples will be collected for additional ctDNA monitoring samples using the Invitae Personalized Cancer MonitoringTM test. Blood samples will be stored at Invitae MetroPark and may be used for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unresectable Pancreatic Cancer
  Interventions: Other: No intervention
- Resectable Pancreatic Cancer
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention associated with this observational study.

SUMMARY:
This is a multicenter, prospective, observational study to evaluate the utility of the Invitae Personalized Cancer MonitoringTM assay for patients with resectable and unresectable pancreatic cancer. Using tumor tissue, a personalized blood test (the Invitae Personalized Cancer MonitoringTM test) will be developed that can be used for repeated monitoring to assess for the presence or absence of circulating tumor DNA (ctDNA). The presence of residual cancer cells after treatment is known as molecular residual disease (MRD) and the detection of ctDNA can provide evidence of the presence of MRD. Participants in this study will have their blood drawn at various time points throughout their cancer treatment to test for ctDNA and monitoring with the Invitae Personalized Cancer MonitoringTM test will continue until disease progression or the duration of the study.

DETAILED DESCRIPTION:
This is a multi-site, prospective, observational trial in Japan of 150 pts with resectable (50) and unresectable (100) PC. The main eligibility criteria are histopathologically diagnosed as adenocarcinoma, no prior treatment for PC, scheduled to undergo surgery for resectable PC or receive systemic therapy for unresectable PC. In resectable PC cohort, blood samples will be collected before surgery and at 1, 3, 6, 9, 12, 18, and 24 months after surgery, and imaging study will be performed before surgery, and at 3, 6, 9, 12, 18, and 24 months after surgery. In the unresectable PC cohort, blood samples will be collected before treatment and at 4, 8, 12, 16, 24, 32, 40, and 48 weeks on treatment, and imaging study will be performed before treatment and every 8 weeks on treatment until 48 weeks. Primary endpoint in the resectable PC cohort is success rate of creating personalized panel using tumor tissue obtained by EUS-FNA/FNB, and that in unresectable PC cohort is rate of concordance of KRAS mutations between tumor tissue and blood samples. Key secondary endpoints in resectable PC cohort are rate of ctDNA positivity for each cancer stage before neoadjuvant chemotherapy and 4 weeks after surgery, and that in unresectable PC cohort is pretreatment ctDNA detection rate for each disease stage.

ELIGIBILITY:
Inclusion Criteria:

A. Unresectable Pancreatic Cancer:

1. At least 20 years of age at the time of consent
2. Histopathologically confirmed adenocarcinoma and diagnosed as having ① or ② described below within 60 days prior to enrollment

   * Clinical Stage Ⅲ (T1-3N2M0, T4 anyNM0)

     * Clinical Stage Ⅳ (anyTanyNM1)
3. Scheduled to receive systemic chemotherapy for unresectable pancreatic cancer.
4. No prior treatment for pancreatic cancer
5. Willing to provide blood and tissue samples in accordance with the research protocol.
6. Adequate tissue samples are available
7. Written informed consent for participating in this study

B. Resectable Pancreatic Cancer:

1. At least 20 years of age at the time of consent.
2. Tissue sample collected by EUS-FNA/FNB and histopathologically diagnosed as having adenocarcinoma.
3. Diagnosed as having cancer meet any one of a to d below within 60 days prior to enrollment

   1. cStage IA (T1 N0 M0)
   2. cStage IB (T2 N0 M0)
   3. cStage IIA (T3 N0 M0)
   4. cStage IIB (T1-3 N1 M0)
4. Scheduled to undergo surgery for resectable pancreatic cancer.
5. No history of prior treatment for pancreatic cancer.
6. Willing to submit blood and tissue samples in accordance with the research protocol.
7. Adequate tissue samples are available
8. Written informed consent for participating in this study

Exclusion Criteria:

Common exclusion criteria for both the unresectable and resectable pancreatic cancer patient cohorts:

1. Synchronous double/multiple cancer or metachronous double/multiple cancer with progression free period of 2 years or shorter.
2. Women who are pregnant or planning to become pregnant.
3. Judged by the investigator as being unsuitable for participation in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with resectable and unresectable Pancreatic Cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cohort of patients with unresectable pancreatic cancer; Rate of concordance of KRAS mutations between tumor tissue and blood samples Primary endpoint | 3 years
  Compare the presence or absence of KRAS mutations in the tumor tissue to the presence or absence of KRAS mutations in the blood for cases in which KRAS is included in the patient specific panel
Cohort of patients with resectable pancreatic cancer; Success rate of WES assays and selections of personalized genes using tumor tissue specimens obtained by EUS-FNA/FNB | 3 years
  Calculate the proportion of patients with resectable pancreatic cancer who are able to successfully have a custom ctDNA panel created with the EUS-FNA/FNB tissue provided

SECONDARY OUTCOMES:
Cohort of patients with unresectable pancreatic cancer; Pretreatment ctDNA detection rate for each disease stage (stage III and stage IV) | 3 years
  Calculate the proportion of patients with stage III and stage IV with a positive Invitae Personalized Cancer Monitoring test prior to receiving any treatment.
Cohort of patients with unresectable pancreatic cancer; Association of pretreatment ctDNA detection rate and the treatment efficacy | 3 years
  Compare the proportion of patients who have a positive versus negative Invitae Personalized Cancer Monitoring test prior to treatment with treatment efficacy as measured by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria after the start of 1st line chemotherapy.
Cohort of patients with unresectable pancreatic cancer; Association of pretreatment serum marker levels (CA19-9) and treatment efficacy | 3 years
  Compare CA19-9 levels in the blood as measured by units per millimeter (u/mL) prior to receiving any treatment to treatment efficacy as measured by RECIST criteria
Cohort of patients with unresectable pancreatic cancer; Association of pretreatment serum marker levels (CEA) and treatment efficacy | 3 years
  Compare CEA levels in the blood as measured by nanograms per milliliter of blood (ng/mL) prior to receiving any treatment to treatment efficacy as measured by RECIST criteria
Cohort of patients with unresectable pancreatic cancer; Association of ctDNA levels and treatment efficacy | 3 years
  Compare ctDNA levels as measured by ctDNA fraction in the Invitae Personalized Cancer Monitoring test prior to receiving any treatment to treatment efficacy as measured by RECIST criteria
Cohort of patients with resectable pancreatic cancer; Rate of ctDNA positivity for each cancer stage (stage IA-stage IIB) before neoadjuvant chemotherapy (NAC) and 4 weeks after surgery | 3 years
  Calculate the proportion of patients by each cancer stage (IA-stage IIB) with a positive Invitae Personalized Cancer MonitoringTM test before the start of neoadjuvant therapy and at the blood draw 4 weeks after surgery.
Cohort of patients with resectable pancreatic cancer; Association of preoperative ctDNA before NAC and overall survival | 3 years
  Compare overall survival between patients who have a positive versus negative Invitae Personalized Cancer MonitoringTM test prior to neoadjuvant treatment
Cohort of patients with resectable pancreatic cancer; Association of postoperative ctDNA before adjuvant chemotherapy (AC) and overall survival | 3 years
  Compare overall survival between patients who have a positive versus negative Invitae Personalized Cancer MonitoringTM test after surgery
Cohort of patients with resectable pancreatic cancer; Proportion of ctDNA positivity at the time of recurrence detected by diagnostic imaging | 3 years
  Calculate the proportion of patients with a positive Invitae Personalized Cancer Monitoring test at the time of clinical recurrence as detected by imaging scans
Cohort of patients with resectable pancreatic cancer, Association of CA-19-9 levels before neoadjuvant chemotherapy and before adjuvant chemotherapy with recurrence free survival | 3 years
  Compare CA19-9 levels as measured by units per millimeter (u/mL) before neoadjuvant chemotherapy and before adjuvant chemotherapy to recurrence free survival
Cohort of patients with resectable pancreatic cancer, association of CEA levels before neoadjuvant chemotherapy and before adjuvant chemotherapy with recurrence free survival | 3 years
  Compare CEA levels as measured by nanograms per milliliter of blood (ng/mL) before neoadjuvant chemotherapy and before adjuvant chemotherapy to recurrence free survival
Cohort of patients with resectable pancreatic cancer, association of ctDNA levels before neoadjuvant chemotherapy and before adjuvant chemotherapy with recurrence free survival | 3 years
  Compare ctDNA levels as measured by ctDNA fraction in the Invitae Personalized Cancer Monitoring test before neoadjuvant chemotherapy and before adjuvant chemotherapy to recurrence free survival
Cohort of patients with resectable pancreatic cancer; Differences in OS and PFS between the patients in whom the personalized panel can be created and those in whom it cannot be created | 3 years
  Compare the ability to generate a personalized ctDNA panel with disease free and overall survival
Cohort of patients with resectable pancreatic cancer; to investigate the lead time of ctDNA detection of recurrence before detection of recurrence via imaging methods | 3 years
  Calculate the lead time as measured by months between a positive Invitae Personalized Cancer Monitoring test and positive imaging findings by either CT or MRI

CONTACTS AND LOCATIONS:
Overall Officials: Taro Shibuki, MD, Principal Investigator — Department of Hepatobiliary and Pancreatic Oncology, National Cancer Center Hospital East, Japan
Locations (1):
- National Cancer Center Hospital East, Kashiwa, Japan